CLINICAL TRIAL: NCT04178954
Title: Semen Analysis and Insight Into Male Infertility
Status: Completed | Type: Observational
Sponsor: Batool Mutar (Other)
Responsible Party: Sponsor-Investigator, Batool Mutar, Prof Dr, Al-Kindy College of Medicine
Organization: Al-Kindy College of Medicine (Other)
Other Study IDs: 11 Al-KindyCM
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2019-12

CONDITIONS: Male Infertility
Keywords: Infertility;; male; semen
MeSH Terms: conditions — Infertility, Male; Infertility

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: semen fluid analysis — semen fluid analysis

SUMMARY:
Semen analysis is the cornerstone for the valuation of the male partner in the infertile couples. This test has been standardized throughout the world through the World Health Organization (WHO) since the1970s by producing, editing, updating, and disseminating a semen analysis manual and guidelines.

DETAILED DESCRIPTION:
A retrospective study to assess the frequency of male factor infertility in the last years.

ELIGIBILITY:
Inclusion Criteria:

* infertile males

Exclusion Criteria:

* suergery

Ages: 15 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: infertile males
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Count and motility | 4 years
  low count

IPD SHARING:
Plan to Share IPD: Undecided